CLINICAL TRIAL: NCT02617368
Title: Fourier Transform of Videokeratography Data: Clinical Usefulness in Moderate and Frome Fruste Keratoconus
Acronym: FFTKC
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Ass. Professor in Ophthalmology, Democritus University of Thrace
Other Study IDs: 304/23/11/2015
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Keratoconus
Keywords: Keratoconus, Corneal crosslinking, Fourier Analysis of Topographic Data
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- KC group: KC group included patients those were diagnosed and classified for moderate keratoconus according to the Amsler-Krumeich classification system
- Forme Fruste Keratoconus Group (FFKG): Forme Fruste Keratoconus Group (FFKG) included patients diagnosed with FFK.
- Control Group (CG): Control group(CG) was formed by refractive surgery candidates.

SUMMARY:
Primary objective of this study was evaluate the diagnostic capacity of fourier analysis of keratometric data in differentiating moderate KC and FFK from healthy corneas.

Study participants were recruited from the Cornea Outpatient service in a consecutive if eligible basis. Two study groups were formed: a)KC group included patients those were diagnosed and classified for moderate keratoconus according to the Amsler-Krumeich classification system, b) FFK group (FFKG) that included patients diagnosed with FFK, and c) Control group (CG) was formed by refractive surgery candidates. Pentacam (Pentacam HR, Oculus Optikgerate GmbH, Heidelberg, Germany)measurements were performed by the same experienced operator in a consistent way.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of keratoconus KC in the fellow eye according to the Amsler-Krumleich criteria (FFKG)
* KISA index between 60 and 100% in the FFK eye (FFKG)
* lack of any KC-related findings / signs in the slit-lamp biomicroscopy (FFKG)
* uneventful ophthalmologic history (CG)
* no indications of corneal pathology in slit-lamp biomicroscopy and Placido *disk-based videokeratography (CG)
* KISA index value less than 60% (CG)
* diagnosed and classified for moderate keratoconus according to the Amsler-Krumeich classification system (KCG)

Exclusion Criteria:

* for all study groups:

  * previous incisional eye surgery
  * corneal scars and opacities
  * history of herpetic keratitis, severe eye dryness
  * pregnancy or nursing
  * current corneal infection
  * glaucoma
  * suspicion for glaucoma
  * IOP lowering treatment
  * underlying autoimmune disease

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants were recruited from the Outpatients Cornea service, in a consecutive if eligible basis
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Spherical Component (SphRmin) | One Day
  Spherical Component (SphRmin) displays the arithmetic mean of all radii of curvature for each ring
Spherical Eccentricity (SphEcc) | One Day
  Spherical Eccentricity is the asphericity that is calculated
Maximum Decentration (MaxDec) | One Day
  decentration or asymmetry of the astigmatic component which is derived from first order component of fourier analysis
Regular Astigmatism at the Center(AstC) | One Day
  the regular astigmatic component is calculated in the center and it is derived from the second order component of Fourier Analysis
Regular Astigmatism at the Periphery (AstP) | One day
  the regular astigmatic component is calculated in the periphery and it is derived from the second order component of Fourier Analysis
Mean Astigmatism (MAst) | One Day
  Mean Astigmatism is the average of astigmatism at the center and the periphery (MAst)
Irregularitiy (Irr) | one Day
Astigmatism at the Center plus the Irregularities (AstCir) | One day
  the irregularities of the cornea which can not be corrected by sphere, cylinder or prism and it is derived from higher order components of Fourier Analysis of Keratometric Data
Total Astigmatism (Tast) which is the sum of Mean Astigmatism and Irregularities. | One Day
  Total Astigmatism (Tast) is the sum of Mean Astigmatism and Irregularities.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute Of Thrace, Alexandroupoli, Evros, Greece